CLINICAL TRIAL: NCT00005191
Title: Clinical Course of Coronary Artery Disease Among Blacks
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1069; R01HL038557 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Heart Diseases

SUMMARY:
To determine the clinical course of coronary artery disease among Blacks receiving medical care for symptomatic heart diseases.

DETAILED DESCRIPTION:
BACKGROUND:

The Black population has age-specific all causes mortality rates among adults which are up to 3.5 times higher than for whites. There remains a pressing need to improve detection and treatment of coronary artery disease among Blacks in an attempt to reduce these unfavorable racial differentials. Also, many fundamental advances in our understanding of atherosclerosis have come from the study of geographic pathology - the epidemiologic comparisons of population groups with widely varying distributions of risk factors. Two prominent features of the epidemiology of coronary artery disease among United States Blacks which are fertile grounds for such comparative studies are the high prevalence of hypertension and the increased susceptibility of Black women to this disease. Knowledge gained from these studies can potentially be applied to coronary artery disease in all human population groups, as has been done with work among the Masai, Seventh-Day Adventists, and other groups.

DESIGN NARRATIVE:

In this longitudinal study, patients were recruited from the adult Emergency Service of Cook County Hospital. Key end-points included: case fatality rates from acute events; long-term survival rates; sudden versus non-sudden death rates; occurrence of first myocardial infarction among patients with new onset angina; functional recovery after myocardial infarction and coronary artery bypass graft. Baseline data were collected in all groups and include: age, sex, education, weight, height, medical history, hyperlipidemia, alcohol and cigarette use, and medications. Both two-dimensional and M-mode echocardiograms were obtained and an exercise test performed. At the time of cardiac catheterization fasting blood samples were drawn for lipid analysis. Bi-plane ventriculography and cineangiography were performed. After discharge, patients returned to the clinic at three-month intervals for up to two years. Analyses were conducted on left ventricular hypertrophy and socioeconomic status as predictors of mortality. The two control groups permitted comparisons of baseline findings and end-points. One hundred and fifty patients from each of the control groups were followed long-term, primarily through surveillance of government vital status records. The study provided data on survival rates, incidence of new events, and mode of death, the roles of sex differences and hypertension in coronary artery disease, and the efficacy of coronary artery bypass surgery.

The study was renewed in FY 1993 to address a series of major questions related to the clinical epidemiology of coronary artery disease among Black women and to continue the on going study involving 2,806 Black men and women who had been enrolled in a hospital-based registry. An examination of the survival patterns and related risk factors in the cohort of 1,559 Black women was the primary focus of this project.

The study was renewed in 1996 to continue to follow the original cohort to examine the interaction of left ventricular hypertrophy (LVH) and mortality risk in the subgroup of patients with coronary heart disease, to investigate further the impact of left ventricular geometry on survival, and to define the prognostic significance of obesity. Also to enroll a new clinical cohort of 5,600 patients, approximately equally divided between Blacks and whites, from Louisiana State University (LSU) Medical Center. The survival patterns of these groups are compared directly, and the contribution of LVH to the Black:white differential estimated. The new cohort serves as a validation sample for the hypotheses derived from the original cohort.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-07; Study Completion 2001-03 (Actual)

REFERENCES:
- [Background] Simmons BE, Castaner A, Santhanam V, Ghali J, Silverman NA, Goldfaden DM, Levitsky S, Cooper R, Ferlinz J. Outcome of coronary artery bypass grafting in black persons. Am J Cardiol. 1987 Mar 1;59(6):547-51. doi: 10.1016/0002-9149(87)91167-2. PMID 3493676
- [Background] Roig E, Castaner A, Simmons B, Patel R, Ford E, Cooper R. In-hospital mortality rates from acute myocardial infarction by race in U.S. hospitals: findings from the National Hospital Discharge Survey. Circulation. 1987 Aug;76(2):280-8. doi: 10.1161/01.cir.76.2.280. PMID 3608117
- [Background] Castaner A, Simmons BE, Mar M, Cooper R. Myocardial infarction among black patients: poor prognosis after hospital discharge. Ann Intern Med. 1988 Jul 1;109(1):33-5. doi: 10.7326/0003-4819-109-1-33. PMID 3377351
- [Background] Ford E, Cooper R, Simmons B, Katz S, Patel R. Sex differences in high density lipoprotein cholesterol in urban blacks. Am J Epidemiol. 1988 Apr;127(4):753-61. doi: 10.1093/oxfordjournals.aje.a114856. PMID 3354542
- [Background] Simmons BE, Castaner A, Campo A, Ferlinz J, Mar M, Cooper R. Coronary artery disease in blacks of lower socioeconomic status: angiographic findings from the Cook County Hospital Heart Disease Registry. Am Heart J. 1988 Jul;116(1 Pt 1):90-7. doi: 10.1016/0002-8703(88)90254-2. PMID 3394636
- [Background] Cooper RS, Simmons BE, Castaner A, Santhanam V, Ghali J, Mar M. Left ventricular hypertrophy is associated with worse survival independent of ventricular function and number of coronary arteries severely narrowed. Am J Cardiol. 1990 Feb 15;65(7):441-5. doi: 10.1016/0002-9149(90)90807-d. PMID 2137665
- [Background] Ghali JK, Liao Y, Cooper RS, Cao G. Changes in pulmonary hemodynamics with aging in a predominantly hypertensive population. Am J Cardiol. 1992 Aug 1;70(3):367-70. doi: 10.1016/0002-9149(92)90621-5. PMID 1632405
- [Background] Liao Y, Cooper RS, Ghali JK, Szocka A. Survival rates with coronary artery disease for black women compared with black men. JAMA. 1992 Oct 14;268(14):1867-71. PMID 1285782
- [Background] Liao Y, Cooper RS, Mensah GA, McGee DL. Left ventricular hypertrophy has a greater impact on survival in women than in men. Circulation. 1995 Aug 15;92(4):805-10. doi: 10.1161/01.cir.92.4.805. PMID 7641360
- [Background] Liao Y, Cooper RS, McGee DL, Mensah GA, Ghali JK. The relative effects of left ventricular hypertrophy, coronary artery disease, and ventricular dysfunction on survival among black adults. JAMA. 1995 May 24-31;273(20):1592-7. PMID 7745772
- [Background] Mensah GA, Barkey NL, Cooper RS. Spectrum of hypertensive target organ damage in Africa: a review of published studies. J Hum Hypertens. 1994 Nov;8(11):799-808. PMID 7853322
- [Background] Fisher SG, Cooper R, Weber L, Liao Y. Psychosocial correlates of chest pain among African-American women. Women Health. 1996;24(3):19-35. doi: 10.1300/j013v24n03_02. PMID 9046551
- [Background] Cooper RS, Liao Y, Rotimi C. Is hypertension more severe among U.S. blacks, or is severe hypertension more common? Ann Epidemiol. 1996 May;6(3):173-80. doi: 10.1016/1047-2797(96)00009-9. PMID 8827151
- [Background] Liao Y, Cooper RS, Durazo-Arvizu R, Mensah GA, Ghali JK. Prediction of mortality risk by different methods of indexation for left ventricular mass. J Am Coll Cardiol. 1997 Mar 1;29(3):641-7. doi: 10.1016/s0735-1097(96)00552-9. PMID 9060905
- [Background] Ghali JK, Liao Y, Cooper RS. Influence of left ventricular geometric patterns on prognosis in patients with or without coronary artery disease. J Am Coll Cardiol. 1998 Jun;31(7):1635-40. doi: 10.1016/s0735-1097(98)00131-4. PMID 9626845
- [Background] Liao Y, Ghali JK, Berzins L, Cooper RS. Coronary angiographic findings in African-American and white patients from a single institution. J Natl Med Assoc. 2001 Dec;93(12):465-74. PMID 11800275